CLINICAL TRIAL: NCT04470726
Title: An Exploratory Study to Evaluate the Safety and Efficacy of AIV001 Intradermally Administered in Subjects With Biopsy-confirmed Basal Cell Carcinoma
Brief Title: Safety and Efficacy Evaluation of AIV001 in Nonmelanoma Skin Cancer of the Low Risk Basal Cell Carcinoma Subtype
Acronym: NMSC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AiViva BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AIV001-C01
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Superficial Basal Cell Carcinoma; Nodular Basal Cell Carcinoma; Nonmelanoma Skin Cancers
Keywords: Nonmelanoma Skin Cancer; Keratinocyte Carcinoma; NMSC; BCC; basal cell carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Intervention Model Description: Subjects will be treated once, twice or three times at 21 days interval and lesions examined at the end of the study investigators will evaluate the lesion surface area for clearance and excise the original lesion area for histological assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AIV001 Treatment Dose 1 (Experimental): Intradermal/intratumoral, Dose 1
  Interventions: Drug: AIV001; Drug: AIV001 suspension
- AIV001 Treatment Dose 2 (Experimental): Intradermal/intratumoral, Dose 2
  Interventions: Drug: AIV001; Drug: AIV001 suspension
- AIV001 Treatment Dose 3 (Experimental): Intradermal/intratumoral, Dose 3
  Interventions: Drug: AIV001; Drug: AIV001 suspension
- AIV001 Treatment Dose 4 (Experimental): Intradermal/intratumoral, Dose 4
  Interventions: Drug: AIV001; Drug: AIV001 suspension

INTERVENTIONS:
Drug: AIV001 — Intradermal/intratumoral
Drug: AIV001 suspension — AIV001 is administered as a aqueous suspension by an intradermal/intratumoral injection

SUMMARY:
To evaluate safety and efficacy of AIV001 treatment on low-risk Nonmelanoma Skin Caner of the basal cell carcinoma subtype.

DETAILED DESCRIPTION:
AIV001 (axitinib) has been formulated to provide focal disease-modifying therapy for patients with nonmelanoma skin cancer (NMSC) of the basal cell carcinoma (BCC) subtype. AIV001 targets angiogenesis, inflammation, and fibrosis associated with various pathological skin conditions and was formulated as a simple intradermal/intratumoral injection demonstrating prolonged skin residence. Surgical excision is the standard treatment for NMSC of the basal cell carcinoma subtype for lesions of < 20 mm. Surgical removal of lesions is effective but for some patients unwilling or contraindicated for surgery a nonsurgical option is needed. A nonsurgical option will eliminate post-surgical complications and scarring experienced after lesion removal. Also, specific anatomical location of lesions present cosmesis (i.e., face) or healing challenges (i.e., lower limbs). An effective injectable will benefit patients who are averse to surgery, at risk of wound healing complications or concerned with cosmesis outcomes or fatigued from multiple surgeries. Patient populations (i.e., elderly or patients with diabetes) who are at risk of delayed wound healing would benefit from an injectable option. This study will evaluate injection methods, interval of treatment, four ascending doses, safety, histological clearance and clinical clearance of biopsy-confirmed "low-risk" BCC lesion of <20 mm located on non-facial skin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 80 years, inclusive
2. No clinically relevant abnormalities identified by a detailed medical history and vital signs
3. Presence of a histologically confirmed low risk BCC lesion, with well-defined borders, and with a largest diameter measure before biopsy of 5 mm to 20 mm, located on arms or trunk
4. Histological diagnosis of the target lesion must have been conducted 5 to 30 days prior to Day 1
5. No other dermatological disease within 50 mm of the target lesion at Day 1
6. No prior or concurrent treatment of the target lesion (including radiation therapy)
7. Willing to undergo surgical excision approximately 63 days after first treatment.

Exclusion Criteria:

1. History or presence of systemic cancer
2. Prior radiation treatment at the lesion site or anywhere else on the body within the past 20 years
3. Concurrent disease or treatment that suppresses the immune system (eg, previous organ transplant history, etc.)
4. Clinically relevant cardiovascular, endocrine, hepatic, neurologic, renal, or other major systemic disease that could complicate execution of the protocol or interpretation of the study results.
5. History of thrombotic events, hemorrhagic events, and gastrointestinal perforation and fistula
6. History of recurrence or presence of any other tumor subtype in the target lesion
7. Concurrent presence of a malignant lesion within 100 mm of the target lesion that will require treatment during the study
8. Current enrollment in any other investigational drug or device study within 60 days of Day 1 of this study
9. Evidence of dermatological disease or confounding dermatological condition that would hinder carrying out the study or interpreting the results (eg, atopic dermatitis, eczema, psoriasis, xeroderma pigmentosa, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Number of adverse events during study period | Approximately 119 days
  Incidence of adverse events
Percentage of Histological Clearance achieved of BCC treated lesion | Cohort 1-3 Day 63; Cohort 4 Day 105 or Day 126
  full clearance is no residual BCC cells by histology

SECONDARY OUTCOMES:
Percentage of Clinical Clearance of treated basal cell carcinoma lesion on skin surface | Cohort 1-3 Day 63; Cohort 4 Day 105 or Day 126
  Number of participants with no surface tumor visible in the study lesion on excision day

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Island Dermatology, Newport Beach, California
  - Skin Surgery Medical Group, San Diego, California
  - Austin Institute for Clinical Research, Pflugerville, Texas